CLINICAL TRIAL: NCT07144332
Title: Assessment of the Efficacy of Hemodialysis on Uric Acid Clearance at End Stage Kidney Disease in Sohag University Hospital
Brief Title: This Study is to Estimate the Efficacy of Hemodialysis Alone for Uric Acid Clearance in Patients on Hemodialysis. In Order to Evaluate the Need of Adjuvant Uric Acid Lowering Therapy
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reham Hussien Abotaleb, Internal medicine resident doctor, Sohag University
Other Study IDs: Soh-Med-25-7-13MS
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Hemodialysis; Hyperuricemia
Keywords: Hemodialysis; Hyperuricemia; chronic kidney disease
MeSH Terms: conditions — Hyperuricemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Uricemia dramatically rises with the stage of chronic kidney disease (CKD) and correlates with its mortality. Hemodialysis (HD) being the most used treatment at the end stage kidney disease in Sohag governorate , we sought to evaluate its efficacy on the clearance of uric acid (UAc) when used alone and twice per week.

Methods: A cross-sectional study of all consenting patients with CKD stage 5 recruited at random during hemodialysis sessions at hemodialysis unit in Sohag university hospital from July to December 2025. We collected socio-demographic data, relevant clinical information, hemodialysis related variables, and measured serum uric acid (SUA) levels before and after the dialysis to assess the uric acid clearance. A clearance between 65 and 80% and above 80% was considered as low and good efficacy of hemodialysis respectively

DETAILED DESCRIPTION:
Aim of the the work The aim of this study is to estimate the efficacy of Hemodialysis alone for uric acid clearance in patients on hemodialysis. In order to evaluate the need of adjuvant uric acid lowering therapy

Patients And Methods

1. Type of The study:

   Prospective cross-sectional study.
2. Place of the study:

   Sohag University Hospital, department of Internal Medicine and hemodialysis unit.
3. Ethical aspect:

Informed Written consent will be taken from all patients to include their data in the study, the research will be approved by medical ethics committee of Faculty of Medicine, Sohag university

Patients:

Inclusion criteria:

• We included all consenting adults aged 18 or older, on maintenance hemodialysis for at least 3 consecutive months receiving 2 to 3 sessions weekly.

Exclusion criteria:

* Patients aged < 18 years old .
* Patients on recent hemodialysis less than 3 months.
* We excluded patients who were on Uric acid lowering therapy (UALT).
* Patients received less than 4 hours of hemodialysis and those who had emergency dialysis.

Number of Patients:

The study will include 100 hemodialysis patients for duration of 6 months.

* Methods We carried out a prospective cross-sectional study at the Hemodialysis unit in Sohag University Hospital . Patients included in the study dialyzed with the Fresenius® 4008S generator (Fresenius Medical Care, St. Wendel, Germany) dialyzers , with a polysulfone synthetic dialysis membrane and bicarbonate dialysate.

The size of the dialysis membrane was estimated according to the total body surface of the patient . Membranes sizes FX60 were used for a body surface of approximately (1.2-1.5 m2 ) ; whereas FX80 between (1.6 and 1.8m2 ) and FX100 were used for body surfaces above 1.8m2.

Dialysis adequacy was calculated from the formula Kt/ V urea; K being the clearance of urea given by the dialyzer, t the duration of the dialysis session (4 h) and V the distribution volume of urea [10].

Uric acid clearance (UAc) was estimated using the formula: UAc=100 x (SUA levels before HD-SUA levels after HD) / SUA levels before HD] [14]. We defined two thresholds values for UAc (65 and 80%).

A Hemodialysis session was considered to be of low efficacy if below 65% of reduction, moderate efficacy between 65 and 80% and a good efficacy above 80% of UAc . [15].

These predictors will be included:

1. Gender.
2. Age.
3. Underlying nephropathy.
4. Average time on renal replacement therapy.
5. Comorbidities,
6. Residual renal function (< 100 ml/24 or ≥ 100 ml/24 h) of participants.
7. Current hemodialysis session parameters such as vascular access.
8. Duration of the session.
9. Time interval between the current and previous dialysis session.
10. Body mass index (BMI).
11. Blood pressure at the beginning and at the end of dialysis
12. Dialysis adequacy.
13. Blood flow (< 300ml/min or>300ml/min).
14. Serum uric acid level which were assessed on a peripheral blood sample collected 5 min before and after dialysis.

Statistical analysis

* All collected data will be analyzed and correlated.
* All the statistical analysis will be done by using Statistical Package for Social Sciences (SPSS Inc., Chicago, IL) version20.
* Baseline data and patient characteristics will be presented using descriptive statistics, for example, number, percentage, mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* We included all consenting adults aged 18 or older, on maintenance hemodialysis for at least 3 consecutive months receiving 2 to 3 sessions weekly

Exclusion Criteria:

1. Patients aged < 18 years old .
2. Patients on recent hemodialysis less than 3 months.
3. We excluded patients who were on Uric acid lowering therapy (UALT).
4. Patients received less than 4 hours of hemodialysis and those who had emergency dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-13 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
study of serum uric acid level in hemodialysis patients | during hemodialysis session 2 to 3 hours
  milligrams per deciliter (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided